CLINICAL TRIAL: NCT00686868
Title: Clinical Phase I/IIA Study of Subcutaneously Administration of Ofatumumab in Rheumatoid Arthritis Patients on Stable Dose Methotrexate
Brief Title: Study to Evaluate SC Route of Administration of Ofatumumab in RA Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OFA110867
Record Dates: First submitted 2008-05-28; First posted 2008-05-30 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Arthritis, Rheumatoid
Keywords: GSK1841157;; rheumatoid arthritis,; B-cell depletion; anti-CD20 monoclonal antibody,
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ofatumumab

STUDY DESIGN:
Who Masked: Participant

ARMS (6):
- 30mg (Experimental): active
  Interventions: Drug: ofatumumab
- 3mg (Experimental): active
  Interventions: Drug: ofatumumab
- 0.3mg (Experimental): active
  Interventions: Drug: ofatumumab
- placebo (Placebo Comparator): placebo
  Interventions: Other: placebo
- 60mg (Experimental): 60mg
  Interventions: Drug: ofatumumab
- 100mg (Experimental): 100mg
  Interventions: Drug: ofatumumab

INTERVENTIONS:
Other: placebo — placebo
  Arms: placebo
Drug: ofatumumab — fully human anti-CD20 monoclonal antibody
  Arms: 0.3mg; 100mg; 30mg; 3mg; 60mg

SUMMARY:
This study will examine the safety and tolerability, PK and PD of subcutaneously administered GSK1841157 in patients with RA on stable dose Methotrexate. The study comprises a single dose escalation/de-escalation phase to investigate the minimal efficacious dose based on PD markers with an acceptable safety profile.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female aged ≥ 18 years
* A diagnosis of rheumatoid arthritis according to the American College of Rheumatology (ACR1987 classification) of at least six months prior to screening
* Subjects must be treated with MTX, 7.5-25 mg/week, for at least 12 weeks prior to Visit 2, with the last 4 weeks prior to Day 2 at a stable dosage
* Patient must be willing to receive folic acid ≥5mg/wk 4 weeks prior to baseline administered according to locally accepted practice
* Body mass index (BMI) < 35kg/m2 (inclusive)
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Key Exclusion Criteria:

* Subjects with a history of a rheumatic autoimmune disease other than RA (except secondary Sjögren's syndrome), or with significant systemic involvement secondary to RA (vasculitis, pulmonary fibrosis or Felty's syndrome)
* Previous exposure to biologic cell depleting anti-rheumatic therapies, including investigational compounds (e.g. anti-CD11a, anti-CD19, anti-CD20, anti-CD22, anti-BLyS/BAFF, anti-CD3, anti-CD4, anti-CD5, anti-CD52)
* Exposure to etanercept < 4 weeks, infliximab or adalimumab < 8 weeks, or abatacept or anakinra < 12 weeks prior to visit 2
* Received any of the following treatments within 4 weeks prior to Visit 2:
* Anti-cancer therapy (e.g. alkylating agents, anti-metabolites, purine analogues, monoclonal antibodies)
* Glucocorticoid unless given in doses equivalent to ≤ 10 mg of prednisolone /day
* Intra-articular, i.m. or IV corticosteroids
* Live/attenuated vaccinations
* Cyclosporine
* Azathioprine
* Penicillamine
* Sulfasalazine
* Bucillamine
* Hydroxychloroquine
* Chloroquine
* Exposure to leflunomide within 12 weeks prior to visit 2 unless the subject has completed peroral cholestyramine treatment
* Exposure to gold therapy ≤ 12 weeks prior to Visit 2
* Exposure to IV immunogammaglobulins ≤ 24 weeks prior to Visit 2
* Past or current malignant melanoma
* Chronic or ongoing active infectious disease requiring systemic treatment such as, but not limited to, renal infection, chest infection with bronchiectasis, tuberculosis and active hepatitis B and C
* History of significant cerebrovascular disease
* Positive plasma / white cell JC Virus (JCV) PCR (either compartment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-06-13 (Actual); Primary Completion 2011-03-11 (Actual); Study Completion 2011-05-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as described by the incidence and severity of adverse events [AEs], clinical laboratory parameters and vital signs. | throughout the study

SECONDARY OUTCOMES:
Requirement for the use of pre-medication, including the timing, type and dose required. | throughout study
Pharmacodynamics (B-cell depletion and re-population) as measured by CD-19 peripheral blood B- lymphocyte count via routine fluorescent activated cell sorting (FACS) analysis. | throughout study
PK/PD parameters including estimation of time to re-population of CD-19 peripheral blood B-cells to above LLQ (and/or <95% depletion) following single subcutaneous dose of Ofatumumab. | throughout study
Immunogenicity as measured by the incidence, titre and type of human anti-human antibody (HAHA) immune response. | throughout study
Other pharmacodynamic/biomarkers of disease activity and immune status may include high sensitivity C-reactive protein (hsCRP), Erythrocyte Sedimentation Rate (ESR), B-Lymphocyte Stimulator (BLyS/BAFF), B-Lymphocyte Chemokine (BLC), IL-6, | throughout study
Immunoglobulins (IgA, IgG, IgM), Complement (CH50, C3, C4), IgM Rheumatoid Factor (IgM-RF), IgA-RF and IgG-RF, anti-cyclic citrullinated peptide antibody (aCCP), | throughout study
serum amyloid A (SAA), CD-3+, CD-4+ and CD-8+ lymphocytes or other biomarkers, as data permit. | throughout study
Pharmacodynamics (B-cell depletion and re-population) as measured by CD-19 peripheral blood B- lymphocyte count via routine FACS analysis.Other Secondary Endpoints | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- United States (2):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Miramar, Florida
- Australia (4):
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Melbourne, Victoria
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Leuven
- GSK Investigational Site, Échirolles, France
- GSK Investigational Site, Verona, Veneto, Italy
- GSK Investigational Site, Christchurch, New Zealand
- GSK Investigational Site, Bydgoszcz, Poland
- Russia (4):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Yaroslavl
- GSK Investigational Site, Madrid, Spain

REFERENCES:
- [Derived] Kurrasch R, Brown JC, Chu M, Craigen J, Overend P, Patel B, Wolfe S, Chang DJ. Subcutaneously administered ofatumumab in rheumatoid arthritis: a phase I/II study of safety, tolerability, pharmacokinetics, and pharmacodynamics. J Rheumatol. 2013 Jul;40(7):1089-96. doi: 10.3899/jrheum.121118. Epub 2013 Jun 1. PMID 23729801
- See also: Results for study OFA110867 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/OFA110867?search=study&search_terms=OFA110867#rs